CLINICAL TRIAL: NCT00149604
Title: Modulation of Visceral Fat by Estrogens After Menopause
Brief Title: AFTER: Altering Fat Through Estrogen and Raloxifene
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG0036; R01AG018198 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Postmenopause
Keywords: metabolic syndrome; hormone therapy; abdominal adiposity; lipolysis
MeSH Terms: conditions — Metabolic Syndrome | interventions — Estrogens, Conjugated (USP); Raloxifene Hydrochloride; Exercise

INTERVENTIONS:
Drug: conjugated estrogens
Drug: Raloxifene
Behavioral: exercise plus mild caloric restriction for weight loss

SUMMARY:
The purpose of this study is to determine whether estrogens specifically promote a reduction in fat from abdominal regions during weight loss and/or prevent the accumulation of abdominal fat during weight gain.

DETAILED DESCRIPTION:
The general aim of this study is to determine whether estrogen-based hormone therapy (HT) in postmenopausal women reduces the accumulation of abdominal visceral fat and whether this is a contributing factor to the effects of estrogens on cardiovascular risk factors. An additional aim is to determine whether raloxifene, a selective estrogen receptor modulator (SERM) that is suggested to be a safer alternative to estrogen for the prevention of osteoporosis, exerts similar effects as estrogen on fat distribution. Mechanisms for possible regional differences in the regulation of fat metabolism in estrogen-sufficient vs estrogen-deficient states will be investigated, as will the extent to which estrogen status and changes in visceral adiposity are associated with changes in risk for coronary artery disease (CAD) and Type 2 diabetes mellitus (DM).

The hypotheses being tested include 1) reductions in total fat mass and total abdominal and visceral fat will be significantly greater in women treated with HT or raloxifene than in those receiving placebo treatment, 2) the accumulation of total fat mass and total abdominal and visceral fat during the 12-month follow-up period will be significantly less in women on HT or raloxifene than in those receiving placebo treatment, 3) a reduction in visceral fat mass will be associated with increased sensitivity to insulin in the breakdown of fat in the whole body, and there will be an independent enhancing effect of HT and raloxifene on insulin action, and 4) changes in risk factors for CAD and Type 2 DM will be more closely associated with changes in visceral adiposity than with changes in total fat mass or other measures of regional adiposity, independent of and in addition to the effects of HT and raloxifene on risk factors.

To meet these aims, a reduction in visceral fat will be induced in 108 postmenopausal women through a 6-month program of supervised exercise training plus mild caloric restriction. Participants will be randomized to receive HT, raloxifene, or placebo. The drug treatment will continue, but the fat reduction program will cease, during a 12-month follow-up period. Risk factors for CAD and Type 2 DM and insulin sensitivity in terms of the breakdown of fat on total body and regional adipose tissue will be evaluated before and after treatment and after the follow-up period (risk factors only). For the purpose of this application, HT refers to a regimen involving daily conjugated estrogens and, in women with a uterus, tri-monthly progestin treatment.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women
* aged 50-70 yr
* healthy, as determined by medical history, physical examination, blood chemistries, and a graded exercise stress test with monitoring of blood pressure and ECG
* good cognitive function.

Exclusion Criteria:

* contraindications to estrogen or raloxifene treatment, including history of or active breast cancer or other estrogen-dependent neoplasms, acute liver disease, undiagnosed vaginal bleeding, and active or history of blood clotting disorders
* mild or more severe cognitive impairment, indicated by a MMSE score <26
* clinically significant abnormal resting electrocardiogram (ECG), angina and/or ECG evidence of acute myocardial ischemia during a maximal exercise stress test
* resting blood pressure above 150 mmHg systolic or 90 mmHg diastolic
* left bundle branch blocks, A-V block greater than first degree, clinically significant arrhythmias
* congestive heart failure
* pulmonary emboli in the previous 6 months
* aortic stenosis
* chronic infections
* orthopedic or other problems that would interfere with participation in the exercise program

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108
Dates: Start 2000-03; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
total body fat mass
total abdominal fat area
visceral abdominal fat area

SECONDARY OUTCOMES:
fat-free mass
total abdominal area
resting metabolic rate
dietary energy intake
cardiovascular fitness
glucose tolerance
blood lipids and lipoproteins
sex hormones (estradiol, estrone, testosterone, sex hormone binding globulin)
glucoregulatory and anti-lipolytic insulin action

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M. Kohrt, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado at Denver and Health Sciences Center, Denver, Colorado, United States

REFERENCES:
- [Background] Espeland MA, Stefanick ML, Kritz-Silverstein D, Fineberg SE, Waclawiw MA, James MK, Greendale GA. Effect of postmenopausal hormone therapy on body weight and waist and hip girths. Postmenopausal Estrogen-Progestin Interventions Study Investigators. J Clin Endocrinol Metab. 1997 May;82(5):1549-56. doi: 10.1210/jcem.82.5.3925. PMID 9141548
- [Background] Margolis KL, Bonds DE, Rodabough RJ, Tinker L, Phillips LS, Allen C, Bassford T, Burke G, Torrens J, Howard BV; Women's Health Initiative Investigators. Effect of oestrogen plus progestin on the incidence of diabetes in postmenopausal women: results from the Women's Health Initiative Hormone Trial. Diabetologia. 2004 Jul;47(7):1175-1187. doi: 10.1007/s00125-004-1448-x. Epub 2004 Jul 14. PMID 15252707
- [Background] Jensen LB, Vestergaard P, Hermann AP, Gram J, Eiken P, Abrahamsen B, Brot C, Kolthoff N, Sorensen OH, Beck-Nielsen H, Nielsen SP, Charles P, Mosekilde L. Hormone replacement therapy dissociates fat mass and bone mass, and tends to reduce weight gain in early postmenopausal women: a randomized controlled 5-year clinical trial of the Danish Osteoporosis Prevention Study. J Bone Miner Res. 2003 Feb;18(2):333-42. doi: 10.1359/jbmr.2003.18.2.333. PMID 12568411
- [Background] Mattiasson I, Rendell M, Tornquist C, Jeppsson S, Hulthen UL. Effects of estrogen replacement therapy on abdominal fat compartments as related to glucose and lipid metabolism in early postmenopausal women. Horm Metab Res. 2002 Oct;34(10):583-8. doi: 10.1055/s-2002-35420. PMID 12439787